CLINICAL TRIAL: NCT00684905
Title: Phase II Interstitial Brachytherapy Combined With Androgen Deprivation Therapy for Locally Recurrent Prostate Cancer After Prior External Beam Irradiation
Brief Title: Leuprolide, Bicalutamide, and Implant Radiation Therapy in Treating Patients With Locally Recurrent Prostate Cancer After External-Beam Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: William Wailing Wong, M.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: 07-00; P30CA015083 (NIH); 7-00 (Other: Mayo Clinic Cancer Center); 7-00 (Other: Mayo Clinic IRB); NCT00956995 (obsolete NCT alias)
Record Dates: First submitted 2008-05-14; First posted 2008-05-28 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Leuprolide; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bicalutamide
Drug: leuprolide acetate
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: quality-of-life assessment
Radiation: brachytherapy

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as leuprolide and bicalutamide, may lessen the amount of androgens made by the body. Implant radiation therapy kills tumor cells by placing material such as radioactive iodine directly into or near a tumor. Giving leuprolide and bicalutamide together with implant radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving leuprolide and bicalutamide together with implant radiation therapy and to see how well it works in treating patients with locally recurrent prostate cancer after external-beam radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and patient tolerance of interstitial brachytherapy combined with androgen-deprivation therapy for patients with locally recurrent prostate cancer after prior external-beam irradiation.
* Determine the toxicity of interstitial brachytherapy combined with androgen-deprivation therapy in these patients.
* Determine the tumor response to interstitial brachytherapy combined with androgen-deprivation therapy in these patients.

OUTLINE: Patients receive neoadjuvant therapy comprising leuprolide acetate intramuscularly for 3 months and oral bicalutamide once daily for 30 days, beginning on the first day of leuprolide acetate administration. Patients then undergo interstitial brachytherapy implantation with I-125. Following brachytherapy, patients receive adjuvant leuprolide acetate every 3 months for an additional 6 months.

Quality of life is assessed at baseline and at every treatment and follow-up visit.

After completion of study therapy, patients are followed every 3 months for 2 years, every to 4-6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven adenocarcinoma of the prostate

  * Locally recurrent disease, defined by digital rectal examination and/or rising prostate-specific antigen (PSA)
* No evidence of nodal or distant metastasis (i.e., N0, M0) on physical examination, bone scan, or CT scan of the pelvis
* Clinical stage T1c-T3a disease at the time of recurrence
* PSA < 10 ng/mL
* Prostate volume by transrectal ultrasonography < 60 cc
* Received prior external beam radiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC ≥ 3,000/μL
* Platelet count ≥ 90,000/μL
* Hemoglobin ≥ 10 g/dL
* Alkaline phosphatase < 2 times normal
* AST < 2 times normal
* Normal prothrombin time and partial thromboplastin time
* No significant obstructive urinary symptoms (AUA score ≤ 16)
* No contraindication for general anesthesia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior transurethral resection of the prostate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2000-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Feasibility
Patient tolerance
Toxicities
Tumor response

CONTACTS AND LOCATIONS:
Overall Officials: William W. Wong, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States